CLINICAL TRIAL: NCT05714852
Title: Promotion of Healthy Eating Behaviors in Type 2 Diabetes Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Valencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Valencia Hospital Clínico
Record Dates: First submitted 2023-01-26; First posted 2023-02-06 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-01

CONDITIONS: Healthy Lifestyle; Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Diet, Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Behavioral: Healthy eating
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Healthy eating — Promotion of healthy eating
  Arms: Intervention

SUMMARY:
Intervention designed to promote healthy eating in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Age
* Type 2 diabetes
* Poor dietary habits

Exclusion Criteria:

* Micro and macro-vascular complications
* Poor glycemic control
* Food allergy

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2025-02-10 (Estimated); Study Completion 2026-02-10 (Estimated)

PRIMARY OUTCOMES:
Change in plasma triglycerides | Before - 16 weeks
  Plasma triglycerides (mmol/L) assessed using chemistry kits on an analyzer platform
Change in blood glucose | Before - 16 weeks
  Plasma blood glucose (mmol/L) assessed using chemistry kits on an analyzer platform

SECONDARY OUTCOMES:
Change in waist circumference | Before - 16 weeks
  Waist circumference in cm assessed using steel tape

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital valencia, Valencia, Spain